CLINICAL TRIAL: NCT01335178
Title: A Program to Protect Young Children From Tobacco Smoke Exposure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Laura Rosen, Chair, Dept. of Health Promotion, School of Public Health, Sackler Faculty of Medicine, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FAMRI-072086_YCSA
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Child Exposure to Tobacco Smoke
Keywords: Tobacco smoke exposure; Secondhand smoke exposure; Passive smoking; Child health; Prevention; Tobacco control; Motivational Interviewing; Air quality; Pilot Study
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Participants received the behavioral intervention, which was designed to motivate parents to protect their children from tobacco smoke exposure
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The intervention consisted of the following elements: (a) Three motivational interviews, scheduled for baseline, one month, and three months; (b) Feedback on air quality in the home (PM2.5 was measured using a Sidepak and/or a Dylos monitoring device, and air nicotine was measured using passive air nicotine dosimeters); (c) Feedback on child's exposure via hair nicotine; (d) a website designed especially for the project [parents.org.il];and (e) various self-help materials, including a booklet, a magnet about TSE, and air fresheners.

SUMMARY:
The goal of this research project is to develop and evaluate an intervention to reduce young child tobacco smoke exposure

DETAILED DESCRIPTION:
Goals The primary goal of this research is to develop and test a theory-based intervention which will reduce tobacco smoke exposure (TSE) of young children. A secondary goal is to increase knowledge of measurement of TSE in young children, and explore the relationship between early TSE, illness, and health care utilization. The study is being conducted in several stages: Developmental (Phase I), Pilot (Phase II), and Trial (Phase III). This registration pertains to Phase II of this trial.

Developmental Stage (Phase I)

This stage includes the following: Systematic reviews of the literature on the topics of encouraging i. parental cessation, ii.reducing child tobacco smoke exposure (TSE), and iii.reducing tobacco smoke air pollution in homes; consultations with experts worldwide; conduct of interviews with parents (n=65) and professionals (n=15) to understand parental perceptions of tobacco smoke exposure, and barriers to protection of children from TSE; and development of an initial intervention program. This stage draws on a social marketing approach and employs in-depth interviews to identify barriers to behavior change and relevant behavior-change recommendations, tailored to the intervention population, and to test the acceptability of program components.

Intervention Program

The intervention consisted of the following elements: (a) Three motivational interviews, scheduled for baseline, one month, and three months; (b) Feedback on air quality in the home (from a Sidepak and/or a Dylos monitoring device, and from passive air nicotine dosimeters); (c) Feedback on child's exposure via hair samples analyzed for nicotine; (d) a website designed especially for the project [22];and (e) various self-help materials, including a booklet, a magnet about TSE, and air fresheners.

Pilot (Phase II) A pilot of the planned intervention was conducted with 29 families. A before - and - after design was used, without a control group. The main endpoint was child exposure to tobacco smoke as measured by hair nicotine. Secondary endpoints included child exposure to tobacco smoke as measured by parental reports, family smoking in home or car, home air nicotine, child illnesses, and use of health services.

[Randomized Controlled Trial (Phase III) (Note: a separate registration number is being sought for this phase) The investigators plan to implement and evaluate the intervention using a randomized controlled trial with an estimated 120 participants. The primary response variable will be child tobacco smoke exposure as measured by hair nicotine. The control group will be offered the intervention at the end of the study (eg, a randomize-to-wait-list design). ]

An effective program for child tobacco smoke exposure reduction could serve as a prototype for reducing child tobacco smoke exposure.

ELIGIBILITY:
Inclusion Criteria:

At least one parent was a current smoker. The child was of the appropriate age (<8 years of age). The child had sufficient hair growth for hair samples. A parent gave consent for participation in the research. The parent can communicate in Hebrew.

Exclusion Criteria:

* One of above conditions not met

Max Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Child exposure to tobacco smoke - hair nicotine | Baseline, 6 months post-intervention
  Child exposure to tobacco smoke as assessed by hair nicotine level

SECONDARY OUTCOMES:
Child exposure to tobacco smoke - parental report | Baseline, 6 months post-intervention
  Child exposure to tobacco smoke as measured by parental report
Child health status | Baseline, 6 months post-intervention (continuous)
  Incidence of respiratory events as reported by parents
Respirable Small Particle (RSPs - PM2.5) level in home | Baseline, 1 month post-intervention
  Measurement of RSPs in the home over a 24-hour period
Air nicotine | Baseline, 6 months post-intervention
  Passive nicotine dosimeters were used for 1 7-day period in the home

CONTACTS AND LOCATIONS:
Overall Officials: Laura J Rosen, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Ramat Aviv, Israel, Israel

REFERENCES:
- [Background] Rosen LJ, Guttman N, Hovell MF, Noach MB, Winickoff JP, Tchernokovski S, Rosenblum JK, Rubenstein U, Seidmann V, Vardavas CI, Klepeis NE, Zucker DM. Development, design, and conceptual issues of project zero exposure: A program to protect young children from tobacco smoke exposure. BMC Public Health. 2011 Jun 28;11:508. doi: 10.1186/1471-2458-11-508. PMID 21711530
- [Result] Rosen LJ, Noach MB, Winickoff JP, Hovell MF. Parental smoking cessation to protect young children: a systematic review and meta-analysis. Pediatrics. 2012 Jan;129(1):141-52. doi: 10.1542/peds.2010-3209. Epub 2011 Dec 26. PMID 22201152
- [Result] Rosen LJ, Myers V, Hovell M, Zucker D, Ben Noach M. Meta-analysis of parental protection of children from tobacco smoke exposure. Pediatrics. 2014 Apr;133(4):698-714. doi: 10.1542/peds.2013-0958. Epub 2014 Mar 24. PMID 24664094
- [Result] Rosen LJ, Tillinger E, Guttman N, Rosenblat S, Zucker DM, Stillman F, Myers V. Parental receptivity to child biomarker testing for tobacco smoke exposure: A qualitative study. Patient Educ Couns. 2015 Nov;98(11):1439-45. doi: 10.1016/j.pec.2015.05.023. Epub 2015 Jun 9. PMID 26160037
- [Result] Rosen L, Zucker D, Hovell M, Brown N, Ram A, Myers V. Feasibility of Measuring Tobacco Smoke Air Pollution in Homes: Report from a Pilot Study. Int J Environ Res Public Health. 2015 Nov 30;12(12):15129-42. doi: 10.3390/ijerph121214970. PMID 26633440
- [Derived] Rosen L, Guttman N, Myers V, Brown N, Ram A, Hovell M, Breysse P, Rule A, Berkovitch M, Zucker D. Protecting Young Children From Tobacco Smoke Exposure: A Pilot Study of Project Zero Exposure. Pediatrics. 2018 Jan;141(Suppl 1):S107-S117. doi: 10.1542/peds.2017-1026N. PMID 29292311
- [Derived] Rosen LJ, Lev E, Guttman N, Tillinger E, Rosenblat S, Zucker DM, Myers V. Parental Perceptions and Misconceptions of Child Tobacco Smoke Exposure. Nicotine Tob Res. 2018 Sep 25;20(11):1369-1377. doi: 10.1093/ntr/ntx169. PMID 29059387